CLINICAL TRIAL: NCT06068816
Title: The Effect of 12 Weeks of Nutritional Supplementation on Nutritional Intake and Status in Older Outpatients With Malnutrition Risk
Brief Title: Effect of Nutritional Supplementation on Nutritional Status & Rehospitalization in Malnourished Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Wageningen University (Other); FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Siti Setiati, Professor of Geriatric Medicine, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Prolansia01
Record Dates: First submitted 2022-03-09; First posted 2023-10-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Malnutrition
Keywords: Malnutrition; Geriatric; Oral nutritional supplement
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to the treatment. Subjects will receive either standard care or standard care plus nutrients dense drinks. Randomization will be done by a third party who is not involved in the study.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessment will be performed by blinded raters.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrient Dense Drink (Experimental): Experimental: Nutrient-dense drink Nutrient-dense drink on top of standard care
  * 200 kcal
  * 15 grams of (whey) protein, 8 grams of fat, and 17 grams of carbohydrates including only 0.2 g lactose
  * 400 IU vitamin D, 250 mg Ca, 10-20 % of the other vitamins/minerals
  Servings :
  • 100 ml water for dissolving 46 g of the served powder
  Interventions: Dietary Supplement: Nutrient-dense drink
- Standard Care (No Intervention): Standard care comprising:
  Standard care only will be provided nutritional counseling to achieve a better nutritional state

INTERVENTIONS:
Dietary Supplement: Nutrient-dense drink — a nutrient-dense drink developed by FrieslandCampina in line with the European Society for Clinical Nutrition and Metabolism guidelines for the dietary management of older malnourished patients
  Arms: Nutrient Dense Drink

SUMMARY:
The primary outcome is the mean difference in energy and protein as well as a selection of micronutrients (calcium, vitamin D, and Vitamin B12) after 12 weeks of intervention between standard care plus nutritional supplementation vs standard care.

The secondary outcomes are body weight, nutritional status, body composition, physical performance, vitamin D level, and nonelective hospitalization

The Study Hypothesize:

The hypothesize that outpatients who receive nutrient-dense drinks (NDD) will have increased body weight, better nutritional status, better body composition, higher vitamin D level, better physical performance and reduced non-elective hospitalization than those receiving standard care after 12 weeks of intervention.

DETAILED DESCRIPTION:
1. Study Design: Randomized Controlled Trial, Randomized and controlled intervention trial with 2 treatments in parallel

   1. Treatment 1: nutrient-dense drinks on top of standard care
   2. Treatment 2: standard care only (reference)
2. Location and time study: Geriatric outpatient clinic and internal medicine outpatient clinic in Cipto Mangunkusumo National Hospital Jakarta. The study will be conducted on July 2022 to October 2023.
3. Study subject: elderly outpatients (aged 60 years old or more) who visit outpatient clinics will be screened for their eligibility as participants of this study.
4. Sample Size: sample size for each group is 41 participants per group (for two groups a total of 82 participants). To anticipate a dropout of 20% a minimum of 98 participants (rounded to 100 participants in total) is the minimum sample size of our study.
5. Data collection : Energy and nutrient intake, particularly protein calcium, vitamin D, and vitamin B12, Nutritional status based on full form Mini Nutritional Assessment, Vitamin D level, lean body mass (using Bioelectrical Impedance Analysis), physical performance will be measured by Shor Physical Performance Battery, handgrip strength, medical history, data on the demographic status and clinical data will be retrieved from the medical record and the attending physicians, body weight and anthropometric measurements, intervention: Nutrient Dense-Drink + Standard Care

ELIGIBILITY:
Inclusion Criteria:

* older patients (60-years or older)
* Malnourished or at risk of malnourished (based on Mini Nutritional Assessment score)

Exclusion Criteria:

* Impaired kidney function (eGFR less than 30 ml/min/1.73 m2)
* Unwillingness to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Changes of Energy in Kilocalories | at baseline and week 12
  Dietary intake will be measured using 3-day dietary food records, 2 weekdays and 1 weekend day)
Changes in Protein intake in grams | at baseline and week 12
  Dietary intake will be measured using 3-day dietary food records, 2 weekdays and 1 weekend day)
Changes in Fat intake in grams | at baseline and week 12
  Dietary intake will be measured using 3-day dietary food records, 2 weekdays and 1 weekend day)
Changes in carbohydrate intake in grams | at baseline and week 12
  Dietary intake will be measured using 3-day dietary food records, 2 weekdays and 1 weekend day)
Changes in micronutrients intake in micrograms | at baseline and week 12
  Dietary intake will be measured using 3-day dietary food records, 2 weekdays and 1 weekend day)

SECONDARY OUTCOMES:
Changes of Mini Nutritional Status Score | at screening (Week 0) and week 12
  The nutritional status will be measured by full form mini nutritional assessment, individuals can be divided in 3 groups using threshold values of <17 for malnourished, 17-23,5 for at risk of malnutrition and ≥ 24 for normal nutritional status with a maximum total score of 30 points
Changes of Vitamin D level | Screening (Week 0) and week 12
  Vitamin D level as a parameter of nutritional status will be measured by the direct competitive chemiluminescence microparticle immunoassay (CMIA) method
Changes of Body Weight | Screening (week 0) and Week 12
  Body weight will be measured in the fasted state to the nearest 0.1 kg with a calibrated digital scale
Changes of Skeletal Muscle Mass | Screening (Week 0) and week 12
  Skeletal Muscle mass will be measured by Bioelectrical Impedance Analysis (BIA) recorded in Kg
Changes of Short Physical Performance Battery Score | Screening (Week 0) and week 12
  Physical performance will be measured by Short Physical Performance Battery, which is measured by scores from Gait speed, chair stand test, and balance test
  Scoring for complete Short Physical Performance Battery
  Category Scores :
  0 - 6 points : poor performance 7-9 points : moderate performance 10-12 points : good performances
Changes of Handgrip Strength | Screening (Week 0) and week 12
  Handgrip strength will be measured by a handgrip dynamometer (recorded in Kg)
Number of the Participants with Rehospitalization | 3 months (12 weeks)
  Non-elective hospitalization will be recorded by medical history
Gait Speed | Screening (Week 0) and week 12
  Outcome recorded in seconds for Baseline, and the Changes (Delta) in 12 weeks
  Additionally, results will be converted into score, which will be used for final SPPB scoring
  3 meter walk: The score is, If time is more than 6''52 sec : 1 point If time is 4"66 to 6"52 sec : 2 points If time is 3"62 to 4"65 sec: 3 points If time is less than 3"62 sec:4 points
Changes to Chair Stand Test | Screening (Week 0) and week 12
  Outcome recorded in seconds for Baseline, and the Changes (Delta) in 12 weeks
  Additionally, results will be converted into score, which will be used for final SPPB scoring
  Participant unable to complete 5 chair stands or completes stands in >60 sec : 0 points If chair stand time is 16"70 sec or more: 1 points If chair stand time is 13"70 to 16"69 sec: 2 points If chair stand time is 11"20 to 13"69 sec: 3 points If chair stand time is 11"19 sec or less: 4 points
  Score will be used for final SPPB scoring

OTHER OUTCOMES:
Balance Test | Screening (Week 0) and week 12
  Outcome recorded in seconds
  A. Side-by-side-stand
  Held for 10 sec ❒ 1 point If participant did not attempt test or failed, circle why:
  Not held for 10 sec ❒ 0 points Tried but unable 1 Not attempted ❒ 0 points Participant could not hold position unassisted 2 If 0 points, end Balance Tests Number of seconds held if instructions less than 10 sec: . sec
  B. Semi-Tandem Stand Held for 10 sec ❒ 1 point Not held for 10 sec ❒ 0 points Not attempted ❒ 0 points (circle reason above) If 0 points, end Balance Tests Number of seconds held if less than 10 sec: . sec
  C. Tandem Stand Held for 10 sec ❒ 2 points Held for 3 to 9.99 sec ❒ 1 point Held for < than 3 sec ❒ 0 points Not attempted ❒ 0 points (circle reason above) Number of seconds held if less than 10 sec: . sec
  Not reported as Secondary outcome but results will be used to calculate SPPB score

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Siti Setiati, MD (Internist Geriatrician),PhD, Principal Investigator — Indonesia University; Prof.Dr.Ing. Lisette CPGM de Groot, PhD, Study Chair — Wageningen University the Netherlands; Esthika Dewiasty, MD (Internist Geriatrician), MSc, Study Director — Universitas Indonesia, PhD candidate at Wageningen University; Sjors Verlaan, PhD, Study Director — FrieslandCampina; Rahmi Istanti, BSc, MPH, Study Director — Indonesia University
Locations (2):
- Indonesia (2):
  - Cipto Mangunkusumo National Hospital, Jakarta
  - Comprehensive Geriatric Clinic, Cipto Mangunkusumo Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: No
All findings of this study will be published in an international open-access journal. Please contact us if any researchers need our individual participant data.